CLINICAL TRIAL: NCT05854043
Title: Modified Enhanced Recovery After Oblique Lateral Interbody Fusion Surgery: a Randomised Controlled Trial
Brief Title: Modified Enhanced Recovery After Oblique Lateral Interbody Fusion Surgery
Acronym: MERAOLIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: xuanwuOLIF
Record Dates: First submitted 2023-04-12; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-04

CONDITIONS: Lumbar Spondylosis; Lumbar Spinal Stenosis; Lumbar Disc Herniation
MeSH Terms: conditions — Spondylosis; Spinal Stenosis; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): In this group, patients will be treated with modified ERAS protocol.
  Interventions: Other: Modified ERAS protocol
- control group (Other): In this group, patients will be treated with routine protocol.
  Interventions: Other: routine protocol

INTERVENTIONS:
Other: Modified ERAS protocol — Modified ERAS protocol for OLIF mainly include perioperative analgesic drug management, operation optimization in the anesthetic management, management of gastrointestinal function, and early mobilization management.
  Perioperative analgesic usage:
  Nonsteroidal anti-inflammatory drugs (NSAIDs) given when Visual Analogue Scale (VAS)>3. Prehabilitation: Respiratory function exercise; walk at least 200 meters daily. Gastrointestinal function management: Oral lactulose use routinely. Sedation and analgesia: patient status index (PSI) 25-50; analgesia nociception index (ANI) 50-70. Local anesthetic: local infiltration around the psoas muscle. Postop off-bed activity: start mobilization within 24h.
  Arms: ERAS group
Other: routine protocol — Perioperative analgesic usage: NSAIDs given follow the patients requirement. Prehabilitation: None. Gastrointestinal function management: None. Sedation and analgesia: bispectral index (BIS) 40-60. Local anesthetic: None. Postop off-bed activity: mobilization follow the patients wish.
  Arms: control group

SUMMARY:
The goal of this randomized clinical trial is to investigate whether modified enhanced recovery after surgery (ERAS) in oblique lumbar interbody fusion (OLIF) can shorten the postoperative hospital stay among patients with lumbar degenerative disease.

The main questions it aims to answer are:

Whether ERAS can shorten the postoperative hospital stay. Whether modified ERAS can improve postoperative functional recovery, improve functional score and pain score, reduce hospitalization costs, improve mental state, and improve abdominal indicators, etc.

Participants will be randomized into modified ERAS group, or control group.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

Whether ERAS can shorten the postoperative hospital stay. Whether modified ERAS can improve postoperative functional recovery, improve functional score and pain score, reduce hospitalization costs, improve mental state, and improve abdominal indicators, etc.

Participants will be randomized into modified ERAS group, or control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old;
* Lumbar degenerative diseases that meet the indications of fusion surgery;
* Patients who are suitable for OLIF surgery;
* Patients who have actually completed OLIF surgery;
* The number of fusion segments is less than or equal to two;
* There was no basis for serious diseases of brain, lung, kidney and other important organs, and preoperative American Society of Anesthesiologists (ASA) score was I-III;
* Agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Patients undergoing lumbar fusion surgery due to spinal trauma;
* Patients undergoing lumbar fusion surgery due to spinal tumor resection;
* Revision surgery;
* The number of fused segments is more than 2;
* Simultaneous lumbar fusion via other approaches, such as transforaminal lumbar interbody fusion (TLIF), posterior lumbar interbody fusion (PLIF), anterior lumbar interbody fusion (ALIF), etc.;
* Pregnancy or perinatal period;
* Blood system diseases lead to coagulation dysfunction;
* Combined with other diseases, life expectancy less than 2 years;
* Patients is participating in other clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative hospital stay | From the date of surgery to discharge, assessed up to 1 month
  The length of hospital stay post-operation.

SECONDARY OUTCOMES:
Postoperative functional recovery | From the date of surgery to discharge, assessed up to 1 month
  Evaluate the functional recovery through 6 Minutes Walk Distance. A longer walk distance indicates better functional recovery.
Postoperative pain score | From the date of surgery to 1 year post-operation
  Postoperative VAS at different time points for pain assessment. From 0-10, 0 indicates no pain, 10 indicates the most severe pain.
Postoperative lumbar neurological function assessment | From the date of surgery to 1 year post-operation
  Postoperative Japanese Orthopedics Association (JOA) at different time points for life quality assessment. From 0-29, A lower score indicates more dysfunction.
Postoperative life quality assessment | From the date of surgery to 1 year post-operation
  Postoperative EuroQol-5 Dimensions (EQ-5D) at different time points for life quality assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Wu, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu hospital capital medical university, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No